CLINICAL TRIAL: NCT05300048
Title: A Phase 1b Study of Serabelisib in Combination With an Insulin Suppressing Diet (Study ISD) and With or Without Nab-paclitaxel in Adult Subjects With Advanced Solid Tumors With PIK3CA Mutations With or Without PTEN Loss
Brief Title: Combination of Serabelisib and Insulin Suppressing Diet With or Without Nab-paclitaxel in Subjects With Advanced Solid Tumors With PIK3CA Mutations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Faeth Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SER-ISD1-001
Record Dates: First submitted 2022-01-31; First posted 2022-03-29 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Advanced Solid Tumor; PIK3CA Mutation; PTEN Loss of Function Mutation
Keywords: PIK3CA Mutation; PTEN Loss of Function Mutation
MeSH Terms: interventions — serabelisib; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Cohort 1a - Dose Modification without nab-paclitaxel (Experimental): Subjects with any solid tumor will receive multiple doses of serabelisib administered orally and will consume Insulin Suppressing Diet for up to 12 months
  Interventions: Drug: Serabelisib; Other: Insulin Suppressing Diet
- Cohort 1b - Dose Modification with Nab-Paclitaxel (Experimental): Subjects with endometrial cancer, ovarian clear cell or ovarian endometriod carcinoma will receive multiple doses of serabelisib administered orally and will consume Insulin Suppressing Diet for up to 12 months. In addition, these subjects will receive nab-paclitaxel intravenously weekly.
  Interventions: Drug: Serabelisib; Other: Insulin Suppressing Diet; Drug: Nab paclitaxel
- Cohort 2 - Expansion Colorectal Cancer (Experimental): Subjects will receive dose of serabelisib as determined from Cohort 1a and 1b, and will consume Insulin Suppressing Diet for up to 12 months
  Interventions: Drug: Serabelisib; Other: Insulin Suppressing Diet
- Cohort 3 - Expansion Endometrial Cancer (Experimental): Subjects will receive dose of serabelisib as determined from Cohort 1a and 1b, and will consume Insulin Suppressing Diet for up to 12 months. If results from Cohort 1b show a favorable risk-benefit ratio, nab-paclitaxel will be administered intravenously weekly.
  Interventions: Drug: Serabelisib; Other: Insulin Suppressing Diet; Drug: Nab paclitaxel
- Cohort 4 - Expansion Ovarian Clear Cell or Ovarian Endometrioid Carcinoma (Experimental): Subjects will receive dose of serabelisib as determined from Cohorts 1a and 1b, and will consume Insulin Suppressing Diet for up to 12 months. If results from Cohort 1b show a favorable risk-benefit ratio, nab-paclitaxel will be administered intravenously weekly.
  Interventions: Drug: Serabelisib; Other: Insulin Suppressing Diet; Drug: Nab paclitaxel

INTERVENTIONS:
Drug: Serabelisib — serabelisib administered orally
Other: Insulin Suppressing Diet — 3 meals consumed daily (i.e., breakfast, lunch, dinner) and optional snacks provided dependent on caloric needs
Drug: Nab paclitaxel — nab-paclitaxel administered intravenously weekly
  Arms: Cohort 1b - Dose Modification with Nab-Paclitaxel; Cohort 3 - Expansion Endometrial Cancer; Cohort 4 - Expansion Ovarian Clear Cell or Ovarian Endometrioid Carcinoma

SUMMARY:
This study will evaluate the feasibility of optimizing the safety and tolerability of serabelisib (an investigational PI3K inhibitor) when combined with an ISD and with or without nab-paclitaxel with a goal of reducing side effects and enhancing anticancer activity.

DETAILED DESCRIPTION:
Targeted anticancer drugs have side effects that often result in a poor quality of life, noncompliance, dose decreases, or discontinuation, all of which can affect efficacy. This study will evaluate the feasibility of optimizing the safety and tolerability of serabelisib when combined with an insulin suppressing diet and with or without nab-paclitaxel with a goal of reducing side effects and enhancing anticancer activity.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide written informed consent.
2. Age ≥18 at Visit -1 (screening).
3. Histologically or cytologically confirmed recurrent solid tumors.

   1. Cohort 1a: any extracranial solid tumor (may include EC, ovarian clear cell, or ovarian endometrioid carcinoma if subject is not eligible for nab-paclitaxel in Cohort

      1b)
   2. Cohort 1b: either recurrent or persistent endometrial adenocarcinoma (EC) with the following histologic epithelial cell types: endometrioid adenocarcinoma, serous adenocarcinoma, undifferentiated carcinoma, clear cell adenocarcinoma, mixed epithelial carcinoma, adenocarcinoma not otherwise specified (N.O.S.), mucinous adenocarcinoma, squamous cell carcinoma, transitional cell carcinoma, and carcinosarcoma or; ovarian cancer (OC) with the primary tumor having ≥ 50% clear cell histomorphology or ovarian clear cell or ovarian endometrioid carcinoma.
   3. Cohort 2: adenocarcinoma of the colon or rectum.
   4. Cohort 3: recurrent or persistent endometrial adenocarcinoma with the following histologic epithelial cell types as described for Cohort 1b
   5. Cohort 4: OC primary tumor carcinomas as described for Cohort 1b
4. Tumor must harbor an activating mutation in the PIK3CA gene with or without PTEN loss, either previously documented or determined during screening.
5. Fresh or archival tumor biopsy with sufficient material to be sent to the designated laboratory for PD analyses. For subjects who consent to future research, an additional 5 slides from a surgical specimen or biopsy is required.
6. Cohort 1a - Dose Modification (subjects with any solid tumor): failed, were intolerant of, or ineligible for no more than three prior lines of therapy (LOT) for advanced/metastatic disease or refused SOC therapy.
7. For all cohorts, in the unlikely scenario that a subject refused all available SOC they may proceed with trial. These subjects would be regarded as having 0 prior LOT.
8. Cohorts 1b, 2, 3, and 4 - failed, were intolerant of, ineligible for, or have refused SOC therapy for advanced/metastatic disease (AJCC stage III and IV) and:

   1. Cohort 2 (subjects with colorectal cancer): Have failed no more than two prior LOT for metastatic CRC.
   2. Cohort 1b, and Cohort 3 (subjects with EC): Have no more than three prior chemotherapeutic regimens for management of endometrial carcinoma (neo-adjuvant and/or adjuvant chemotherapy will be counted as one prior LOT). Prior hormonal therapy will not count as a systemic regimen.
   3. Cohort 1b, and Cohort 4 (subjects with clear cell or endometrioid OC): Subjects must have had no more than three prior chemotherapeutic regimens for management of ovarian carcinoma. Prior hormonal therapy will not count as a systemic regimen.
9. Life expectancy of at least 3 months.
10. At least one measurable lesion (as defined by Response Evaluation Criteria in Solid Tumors [RECIST] 1.1).
11. ECOG PS of 0 to 1.
12. Adequate organ function

    1. Absolute neutrophil count (ANC) ≥1.0 × 10^9/L or ≥1.5 x 10^9/L if planned to be treated with nab-paclitaxel, platelet count ≥75 × 10^9/L, and hemoglobin ≥8.5 gm/dL (may be transfused to reach this hemoglobin level unless due to blood loss).
    2. Liver transaminases (AST and ALT) ≤2.5 × upper limit of normal (ULN) (<5 × ULN if liver metastases are present), and total bilirubin ≤1.5 × ULN (<3 x ULN if subject has Gilbert Syndrome).
    3. INR ≤1.5 x ULN unless subject is on anticoagulants that would affect the INR, then INR must be in the desired therapeutic range as judged by the Investigator.
    4. Albumin level ≥3.0 mg/dL or ≥ the lower limit of normal.
    5. Renal: Serum creatinine ≤2 x ULN
13. Ability to take PO medication, be willing to adhere to study procedures and Study Intervention administration, and receive, consume, and comply with Study ISD.
14. For women of child-bearing potential, a negative serum pregnancy test collected at screening (Visit-1) and negative urine pregnancy test collected at baseline (Visit-1) and use of physician-approved method of birth control from the time of the pregnancy test performed at screening to 90 days following the last administration of Study Drug or, if applicable, 6 months following the last administration of nab-paclitaxel.
15. Male subjects must be surgically sterile or must agree to use physician-approved contraception during the study and for 90 days following the last administration of Study Drug.

Exclusion Criteria:

1. Diagnosis of primary malignant brain tumor.
2. Has had serabelisib, alpelisib, or other PI3K inhibitor.
3. Leptomeningeal disease and symptomatic or untreated brain metastases.
4. Diagnosis of, or requiring treatment for, another malignancy within the past 2 years (excluding a history of carcinoma in situ of the cervix, superficial non-melanoma skin cancer, or superficial bladder cancer that has been adequately treated, or stage 1 prostate cancer that does not require treatment or requires only treatment with luteinizing hormone-releasing hormone agonists or antagonists if initiated at least 90 days prior to the first dose of Study Drug).
5. Is less than 21 days from therapeutic radiation or chemotherapy prior to the first day of dosing with Study Drug and has not recovered to Grade ≤ 1 from all clinically significant toxicities related to prior therapies.
6. For subjects receiving nitrosoureas or mitomycin C, the subject is < 6 weeks from last dose. For monoclonal antibody therapy, the subject is < 1 half-life or <4 weeks from the last dose.
7. Chronic, systemically administered glucocorticoids in doses equivalent to >5 mg prednisone daily. Replacement corticosteroids for adrenal insufficiency are permitted.
8. Diabetes mellitus requiring insulin or insulin secretagogue therapy.
9. Poorly controlled diabetes mellitus defined as glycosylated hemoglobin A1c (HbA1c) >7.5% or fasting blood sugar >160 mg/ dL.
10. Known impaired cardiac function or clinically significant cardiac disease.
11. QTcF interval >470 msec found at screening.
12. Myocardial infarction, cardiac stent placement, or unstable angina within 6 months before the first administration of Study Drug.
13. Have clinically significant peripheral vascular disease.
14. Manifestations of malabsorption
15. Other clinically significant comorbidities.
16. Pregnant (positive serum pregnancy test), planning to become pregnant during the study, or breastfeeding/planning to breastfeed during the study.
17. Have taken strong CYP3A4 inducers/inhibitors within 7 days before the first administration of serabelisib or have conditions that require the concomitant use of CYP3A4 inducers/inhibitors.
18. Untreated or poorly controlled, gastro-esophageal reflux disease.
19. Have taken histamine-H2 receptor antagonists within 12 hours before the first administration of serabelisib.
20. Have taken PPI within 7 days or 5 half-lives (whichever is the shorter duration) before the first administration of serabelisib or are anticipated to need PPI during the study.
21. Have taken neutralizing antacids within 4 hours before the first administration of serabelisib or are anticipated to need frequent antacid use during the study.
22. Subjects with poorly controlled human immunodeficiency virus, hepatitis B virus, and/or hepatitis C virus infections.
23. Known allergies to nab-paclitaxel or excipients, serabelisib or excipients or the ISD
24. Severe, uncontrolled gout.
25. A BMI <18.5 kg/m2, or serious or refractive cachexia or anorexia that, in the Investigator's opinion, realistically prohibits subjects from having energy or appetite sufficient to reliably engage in a strict ISD regimen for an extended time.
26. Any condition that renders the subject unable to satisfactorily chew, swallow, digest, or tolerate (i.e., persistent diarrhea) the majority of foods and liquids of the Study ISD.
27. History of severe nephrolithiasis requiring urologic intervention.
28. Participation in a diet or weight loss plan within 10 days prior to the first administration of Study Drug.
29. Severe constipation or condition where exacerbation of constipation is not advisable (eg, small bowel obstruction history).
30. History of anaphylaxis from food allergy or other disease state requiring avoidance of a particular food, such as celiac disease.
31. Diagnosed eating disorder in the past 10 years.
32. Unwilling to take a non-vegan or non-vegetarian diet.
33. Peripheral neuropathy ≥ CTC Grade 2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2022-04-22 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Cohorts 1a/1b: Evaluate safety | Through study completion, up to 12 months.
  Incidence of related AEs
Cohorts 1a/1b: Evaluate compliance | Through study completion, up to 12 months.
  Compliance of Study intervention
Cohorts 1a/1b: Evaluate the pharmacokinetic impact by measuring Cmax. | Through study completion, up to 12 months.
  Standard pharmacokinetic parameters (Cmax)
Cohorts 1a/1b: Evaluate the pharmacokinetic impact by measuring Tmax. | Through study completion, up to 12 months.
  Standard pharmacokinetic parameters (Tmax).
Cohorts 1a/1b: Evaluate the pharmacokinetic impact by measuring AUC. | Through study completion, up to 12 months.
  Standard pharmacokinetic parameters (AUC).
Cohorts 2, 3, 4: Use the Objective Response Rate (ORR) to assess the antitumor efficacy of serabelisib in combination with a Study ISD. | Through study completion, an average of 8 months.
  Proportion of subjects who have best overall response of either complete response (CR) or partial response (PR)

SECONDARY OUTCOMES:
Cohorts 1a/1b: Antitumor efficacy of study intervention by measuring ORR. | Through study completion, up to 12 months.
  Proportion of subjects who have best overall response of either CR or PR, as determined by each site.
Cohorts 1a/1b: Antitumor efficacy of study intervention by measuring PFS. | Through study completion, up to 12 months.
  Time from date of first dose of Study Drug (Visit 1) to the date of first evidence of disease progression or death from any cause (whichever occurs first).
Cohorts 1a/1b: Antitumor efficacy of study intervention by measuring OS. | Through study completion, up to 12 months.
  Overall survival (OS) and landmark survival.
Cohorts 1a/1b: Antitumor efficacy of study intervention by measuring DoR. | Through study completion, up to 12 months.
  Duration of response (DoR)
Cohorts 1a/1b: Antitumor efficacy of study intervention by measuring DCR. | Through study completion, up to 12 months.
  Disease control rate (DCR; CR + PR + stable disease [SD])
Cohort 2, 3, 4: Confirm safety | Through study completion, up to 12 months.
  Incidence of related AEs
Cohort 2, 3, 4: Confirm the compliance of study intervention. | Through study completion, up to 12 months.
  Compliance of Study intervention
Cohort 2, 3, 4: Additional assessments of antitumor efficacy of study intervention (Measuring PFS). | Through study completion, up to 12 months.
  Time from the date of first dose of Study Drug (Visit 1) to the date of first evidence of disease progression or death from any cause (whichever occurs first)
Cohort 2, 3, 4: Additional assessments of antitumor efficacy of study intervention (Measuring OS). | Through study completion, up to 12 months.
  OS and landmark survival
Cohort 2, 3, 4: Additional assessments of antitumor efficacy of study intervention (Measuring DoR). | Through study completion, up to 12 months.
  DoR
Cohort 2, 3, 4: Additional assessments of antitumor efficacy of study intervention (Measuring DCR). | Through study completion, up to 12 months.
  DCR (CR+PR+SD)
Cohort 2, 3, 4: Assess the population PK and intra-tumoral concentration of study intervention. | Through study completion, up to 12 months.
  Standard PK Parameters (Cmax) in plasma.
Cohort 2, 3, 4: Assess the population PK and intra-tumoral concentration of study intervention. | Through study completion, up to 12 months.
  Standard PK Parameters (Tmax) in plasma
Cohort 2, 3, 4: Assess the population PK and intra-tumoral concentration of study intervention. | Through study completion, up to 12 months.
  Standard PK Parameters (AUC) in plasma
Cohort 2, 3, 4: Assess the population PK and intra-tumoral concentration of study intervention. | Through study completion, up to 12 months.
  Serabelisib concentration in tumor tissue

OTHER OUTCOMES:
Cohorts 1a/1b, 2, 3, 4: Assessment of PD of study intervention. | Through study completion, up to 12 months.
  Change in PD markers (insulin)
Cohorts 1a/1b, 2, 3, 4: Assessment of PD of study intervention. | Through study completion, up to 12 months.
  Change in PD markers (glucose)
Cohorts 1a/1b, 2, 3, 4: Assessment of PD of study intervention. | Through study completion, up to 12 months.
  Change in biomarkers of insulin-PI3K signaling
Cohorts 1a/1b, 2, 3, 4: Assessment of PD of study intervention. | Through study completion, up to 12 months.
  Changes in tumor marker levels.
Cohorts 1a/1b, 2, 3, 4: Assessment of immune markers in response to study intervention. | Through study completion, up to 12 months.
  Assessment of immune markers in PBMCs throughout study.
Cohorts 1a/1b, 2, 3, 4: Assessment of genetic predictors of efficacy. | Through study completion, up to 12 months.
  Analysis into whether the genetic status of the patient predicts a positive or negative therapeutic response (efficacy).
Cohorts 1a/1b, 2, 3, 4: Assessment of genetic predictors of toxicity. | Through study completion, up to 12 months.
  Analysis into whether the genetic status of the patient predicts susceptibility to AEs (toxicity).

CONTACTS AND LOCATIONS:
Overall Officials: Vicky Makker, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (17):
- United States (17):
  - University of Alabama, Birmingham, Alabama
  - Pacific Cancer Specialists, Anaheim, California
  - Valkyrie Clinical Trials, Los Angeles, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Community Health Network, Inc., Indianapolis, Indiana
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - New Jersey Cancer Care, PA, Belleville, New Jersey
  - Englewood Health, Englewood, New Jersey
  - Northwell Health, Lake Success, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - East Carolina University, Greenville, North Carolina
  - University of Pennsylvania Health System, Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Baptist Hospitals of Southeast Texas, Beaumont, Texas
  - Oncology Consultants, PA, Houston, Texas
  - Lumi Research, Kingwood, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No